CLINICAL TRIAL: NCT03345316
Title: Safety and Usability Evaluation Study of FFI-1010 Single Administration for Children Under 18 Years Old With Kidney Disease (Phase III Study).
Brief Title: Study of FFI-1010 in Pediatric Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FFI-1010-004
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Children Under 18 Years Old With Kidney Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FFI-1010 (Experimental)
  Interventions: Drug: FFI-1010

INTERVENTIONS:
Drug: FFI-1010 — Intravenous single dosing

SUMMARY:
The purpose of this study is revealing that the ratio of creatinine clearance (Ccr) to inulin clearance (Cin) measuring at the same time is more than 1.2.

ELIGIBILITY:
Inclusion Criteria:

* Kidney disease patients requiring exact evaluation of kidney function
* eGFR: >=30 and <=89 mL/min/1.73m^2

Exclusion Criteria:

* Edema on the day before start of study treatment
* Oliguria on the day before start of study treatment
* Dehydration on the day before start of study treatment
* Infection or inflammatory disease before administration
* History of epilepsy or organic brain disorder
* History of, clinically significant cardiac, hematologic, hepatic and pancreatic disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Ratio of Cin to Ccr measuring at the same time | 120 minutes
  Demonstrating usability of inulin clearance by comparison between inulin clearance and creatinine clearance at the same time after the start of FFI-1010 administration

CONTACTS AND LOCATIONS:
Locations (1):
- Fuji Yakuhin Investigational sites, Tokyo, Japan

REFERENCES:
- [Derived] Uemura O, Ishikura K, Kamei K, Hamada R, Yamamoto M, Gotoh Y, Fujita N, Sakai T, Sano T, Fushimi M, Iijima K. Comparison of inulin clearance with 2-h creatinine clearance in Japanese pediatric patients with renal disease: open-label phase 3 study of inulin. Clin Exp Nephrol. 2022 Feb;26(2):132-139. doi: 10.1007/s10157-021-02133-5. Epub 2021 Sep 25. PMID 34562149